CLINICAL TRIAL: NCT04269668
Title: An Open-label, Two-center, Randomized, Cross-over Study to Evaluate the Safety and Efficacy of Glycemic Control Using Hybrid-closed Loop vs. Advanced Hybrid Closed-loop in Young Subjects With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: GIF (Unknown); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMC077719ctil
Record Dates: First submitted 2020-02-06; First posted 2020-02-17 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Hybrid Closed Loop; Closed Loop; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Medtronic Minimed 670G 3.0 HCL (Active Comparator): Hybrid closed loop system
  Interventions: Device: Medtronic Minimed 670G 3.0 HCL
- Medtronic Minimed 670G 4.0 AHCL (Experimental): Advanced hybrid closed loop system
  Interventions: Device: Medtronic Minimed 670G 4.0 AHCL

INTERVENTIONS:
Device: Medtronic Minimed 670G 3.0 HCL — Hybrid closed loop system
  Arms: Medtronic Minimed 670G 3.0 HCL
Device: Medtronic Minimed 670G 4.0 AHCL — Advanced hybrid closed loop system
  Arms: Medtronic Minimed 670G 4.0 AHCL

SUMMARY:
Closed-loop systems are becoming an integral part of diabetes management. These systems were uniformly proven to improve glycemic control, reduce hyperglycemia and hypoglycemia while modestly reducing HbA1c levels and improving quality of life. While overnight control is close to optimal under closed loop control, postprandial hyperglycemia during daytime remains a challenge. The advanced hybrid closed loop system was designed with an improved auto-basal control and additional auto-bolus module that delivers correction boluses automatically. In addition, this system was developed to improve user experience by significantly reducing the amount of alarms and exits from Auto Mode. Therefore, this system might have an advance in treating hyperglycemia over the hybrid closed loop that controls glucose levels by modulation of insulin basal rate only. Therefore, we propose the current study that will compare 6 weeks glycemic control using hybrid closed loop versus advanced hybrid closed loop that add correction boluses among young children and adolescents.

The objective of this study is to evaluate and compare the safety and efficacy of 6 weeks glucose control using Hybrid Closed Loop (HCL-670G) compared to Advanced Hybrid Closed Loop System (AHCL- 670G) in young subjects with sub-optimally controlled type 1 diabetes. A total of 28 subjects (age 7-14 years) will be enrolled at two investigational centers.

At the end of the cross-over study participants will be offered with an extension period, during which they will be offered to use their preferred closed-loop system for another 3 months

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1 duration >1 year since diagnosis
* Pump therapy for at least 3 months and experience with sensor use
* Age >=7 years up to 14 years
* A1C>7.5% and <10.0%
* BMI SDS below the 95th percentile for age
* Subjects who live with at least one other adult person, who will be trained in managing an emergent hypoglycemia and who is able to contact the study subject any time
* Subjects/caregivers capable of operating a computer-based system

Exclusion Criteria:

* Subject is unable to tolerate tape adhesive in the area of sensor placement
* Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
* Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study drug or device in the last 2 weeks
* Subject has a positive pregnancy screening test
* Subject is female, sexually active without the use of contraception, and plans/able to become pregnant during the course of the study and is not using an acceptable method of contraception or breast feeding women
* Subject has had hypoglycemia resulting in loss of consciousness with or without seizure within the past 6 months prior to screening visit
* Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to screening visit
* Subject has a history of a seizure disorder
* Subject has central nervous system or cardiac disorder resulting in syncope
* Subject has eating disorder
* Subjects with a history of adrenal insufficiency or chronic renal diseases
* Subjects with history of migraines that have occurred at least 2 times in the last 3 months prior to enrollment
* Any disease or condition that may influence the A1C testing e.g. abnormal red blood cell indices and iron deficiency, sickle cell disease, hemoglobinopathy
* Subject needs to travel by air during the study duration
* Medication influencing coagulation as Marcumar or systemic Xa-Antagonists -Untreated coeliac disease (Transglutaminase in the last 6 months elevated 2x>upper limit)
* Mental incapacity or psychiatric disorders (Major Depression, anxiety disorders, schizophrenia)
* Coagulation disorder, wound healing disorder
* Severe diseases as cancer, heart failure, M. Parkinson, M. Addison, hyper or hypothyroidism, diabetic nephropathy or neuropathy or cardiomyopathy
* Patients with Diabetes mellitus Type 2
* Patients not willing to perform at least 4 blood glucose measurements a day.
* Patients with a need of less than 8 IUE or more than 250 IUE a day.
* Patients who are not willing to or not able to stay in contact with their physician.
* Patient abusing illicit drugs, prescription drugs or alcohol
* Patient is using other (other than insulin) diabetic medication incl. pramlintide (Symlin) DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors).
* Patient or caregiver are expected to be incompliant with study procedures or instructions (e.g. sensor change, using the bolus wizard, falsifying carbohydrate intake) or are unlikely to understand study procedures or instructions.
* Patient takes any oral, injectable, or IV steroids (incl. glucocorticoids).
* Patients whose health or safety would be compromised by study participation according to the investigator's judgement.
* Patient is taking any medication that is a contraindication for study participation according to the discretion of the investigator.
* Patients who may have a risk not to realize acoustic or visual alarms due to visual or hearing impairment.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-07-19 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Percentage of time of glucose sensor readings within 70 to 180 mg/dl | 6 weeks for each arm of the crossover, day 90 of the extension period
Percentage of time of glucose sensor readings below 54 mg/dl | 6 weeks for each arm of the crossover

SECONDARY OUTCOMES:
Percentage of time of glucose levels spent below 70 mg/dl | 6 weeks for each arm of the crossover, day 90 of the extension period
Percentage of time of glucose levels spent above 180 mg/dl | 6 weeks for each arm of the crossover, day 90 of the extension period
Average glucose sensor readings | 6 weeks for each arm of the crossover, day 90 of the extension period
Standard deviation of glucose sensor readings | 6 week for each arm of the crossover, day 90 of the extension period
Fasting blood glucose levels | 6 weeks for each arm of the crossover, day 90 of the extension period
HbA1c change | 6 weeks for each arm of the crossover, day 90 of the extension period
Amount of total insulin delivery | 6 weeks for each arm of the crossover, day 90 of the extension period
Amount of basal insulin delivery | 6 weeks for each arm of the crossover, day 90 of the extension period
Amount of bolus insulin delivery | 6 weeks for each arm of the crossover, day 90 of the extension period
Serious Adverse Events (SAE) | 6 weeks for each arm of the crossover, day 90 of the extension period
Serious Adverse Device Events (SADE) | 6 weeks for each arm of the crossover, day 90 of the extension period
Unanticipated Adverse Device effects (UADE) | 6 weeks for each arm of the crossover, day 90 of the extension period
Incidence of Severe Hypoglycemia | 6 weeks for each arm of the crossover, day 90 of the extension period
incidence of DKA | 6 weeks for each arm of the crossover, day 90 of the extension period

OTHER OUTCOMES:
Percentage of time of glucose sensor readings below 60 mg/dl | 6 weeks for each arm of the crossover
Percentage of time of glucose sensor readings above 250mg/dl | 6 weeks for each arm of the crossover
Percentage of time of glucose sensor readings above 300mg/dl | 6 weeks for each arm of the crossover
percentage of time of using the closed loop system | 6 weeks for each arm of the crossover, day 90 of the extension period
INSPIRE questionnaire measures | 6 weeks for each arm of the crossover, day 90 of the extension period
  The INSPIRE questionnaire measures Insulin delivery System's Perceptions, Ideas, Reflections and Expectations

CONTACTS AND LOCATIONS:
Locations (2):
- Diabetes -Zentrum fuer kinder und jugendliche, Hanover, Germany
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel